CLINICAL TRIAL: NCT05486286
Title: Clinical Study of a Real-time Video-assisted System for Nasogastric Tube Placement
Brief Title: Video Assisted System for Nasogastric Tube Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Chiao-Hsiung Chuang, Associate Professor, National Cheng-Kung University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B-BR-111-006
Record Dates: First submitted 2022-07-26; First posted 2022-08-03 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Enteral Nutrition

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- video assisted NG placement (Experimental): This is a single-arm study. A live-video system (NCKU-NG system) was developed to assist in the placement of enteral feeding tubes.
  Interventions: Device: NCKU-NG system

INTERVENTIONS:
Device: NCKU-NG system — A live-video system (NCKU-NG system) was developed to assist in the placement of enteral feeding tubes. This system consists of a camera and light source that can be inserted into the commercial NG tube to view live video during feeding tube placement. Manual air insufflation may aid feeding tube placement and improve visualization of anatomic landmarks. After the procedure, an abdominal X-ray is done to confirm the position of the feeding tube.

SUMMARY:
A live-video system (NCKU-NG system) was developed to assist in the placement of an enteral feeding tube. This system consists of a camera and light source that can be inserted into the commercial NG tube to view live video during feeding tube placement. Manual air insufflation can be used to aid feeding tube placement and improve visualization of anatomic landmarks. After the procedure, an abdominal X-ray is done to confirm the position of the feeding tube.

DETAILED DESCRIPTION:
This study used 15 Fr feeding tubes with an outer diameter of 4.5 mm and an inner diameter of 3.5 mm (Freka®, Bad Homburg, Germany). Patients were advised to maintain nothing by mouth (NPO) for at least four hours before the placement. An insufflation device (Olympus, Tokyo, Japan) was utilized whenever necessary to facilitate feeding tube placement or confirm its position. In cases where misplacement into the trachea was detected, the feeding tube was carefully withdrawn and reinserted into stomach. After successful insertion, all feeding tubes were securely fixed with tape on the nose. The position of NG tube was reconfirmed by traditional auscultation. Chest X-ray imaging was performed for every patient after the NG tube placement to verify the positioning of the tube by the primary care physician. Time to visual confirmation of stomach position, for completing tube placement with/without air insufflation were recorded. Numbers of attempts, vocal cord/trachea visualization and air insufflation were also recorded. A study assistant monitored the patient's condition for the subsequent seven days, recording any observed complications or adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Patients (>20 y/o) requiring enteral feeding and/or medication with an expected duration longer than 48 hours were eligible for inclusion.

Exclusion Criteria:

* Patients can't receive an X-ray after the procedure to confirm tube position (e.g. pregnancy)
* Patients with hemodynamic instability (defined as mean arterial pressure <65 mmHg)
* Patients with a history of basal skull fracture.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-08-02 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2023-05-10 (Actual)

PRIMARY OUTCOMES:
The successful rate (percent) of gastric placement of feeding tubes | up to 24 hours after chest X-ray
  The successful rate (percent) of gastric placement of feeding tubes using the video-assistance system (NCKU-NG system), was assessed by X-ray.

SECONDARY OUTCOMES:
opearator evaluation (Liker scale) | immediately after procedure
  The operator will evaluate the 1) feasibility of video assistance placement, 2) imaging clearance, 3) whether is it easy to remove the camera probe after reaching the stomach, 4) whether is it easy to confirm the gastric position. All the evaluation is cored on a Liker scale (1-5, whether higher scores mean a better outcome)

OTHER OUTCOMES:
Procedure time needed (minutes) | Immediately after procedure
  The time to insertion of NG tube (from the nose insertion till reaching the stomach)
number of patients with visualization of the trachea (n, %) | immediately after procedure.
  Evaluate how many patient has trachea miss-insertion under this video-assistance

CONTACTS AND LOCATIONS:
Overall Officials: Chiao-Hsiung Chuang, M.D., Principal Investigator — Department of Internal medicine, National Cheng-Kung University Hospital
Locations (1):
- Chuang Chiao-Hsiung, Tainan, Taiwan